CLINICAL TRIAL: NCT03833817
Title: A Communication-based Intervention for Advanced Cancer Patient-caregiver Dyads to Increase Engagement in Advance Care Planning and Reduce Caregiver Burden
Brief Title: Patient-caregiver Communication Intervention for Prognostic Understanding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1803019107; R21CA224874 (NIH)
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Results first posted 2022-08-18 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-07

CONDITIONS: Advanced Cancer
Keywords: advance care planning; prognostic understanding; communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient intervention arm (Experimental): This intervention arm contains the patients from this single arm study in which patients and caregivers will be given the experimental intervention (TAC intervention) with assessments pre and post intervention. The intervention will consist of six 45-minute telephone-delivered sessions. Session topics will include: (a) Distress management/tolerance (Sessions 1 and 2); (b) communication skills (Sessions 3 and 4); (c) guided review of prognostic information (Session 5); and (d) Intervention review and future plan (Session 6). Sessions will be completed by the individual (Sessions 1 and 3) and dyad (Sessions 2, and 4-6).
  Interventions: Behavioral: Talking about Cancer (TAC)
- Caregiver (of patient) intervention arm (Experimental): This intervention arm contains the caregivers of patients from this single arm study in which patients and caregivers will be given the experimental intervention (TAC intervention) with assessments pre and post intervention. The intervention will consist of six 45-minute telephone-delivered sessions. Session topics will include: (a) Distress management/tolerance (Sessions 1 and 2); (b) communication skills (Sessions 3 and 4); (c) guided review of prognostic information (Session 5); and (d) Intervention review and future plan (Session 6). Sessions will be completed by the individual (Sessions 1 and 3) and dyad (Sessions 2, and 4-6).
  Interventions: Behavioral: Talking about Cancer (TAC)

INTERVENTIONS:
Behavioral: Talking about Cancer (TAC) — The TAC intervention is a six session intervention designed to teach the techniques of distress tolerance and communication skills in order to assist patients and their caregivers in discussing the patients' prognoses.

SUMMARY:
The purpose of this study is to: (1) develop a communication-based intervention to improve advanced cancer patients' and caregivers' prognostic understanding using communication strategies (e.g., acknowledgment, validation of fears) and distress management techniques (e.g., deep breathing, muscle relaxation); (2) evaluate the feasibility and acceptability of the intervention among advanced cancer patients and their caregivers; and (3) test the preliminary efficacy of the intervention on patients' and caregivers' prognostic understanding (primary outcome); completion of DNR order, living will, and health care proxy; psychological distress; communication quality; caregiver burden; and healthcare utilization (secondary outcomes).

ELIGIBILITY:
Patient Inclusion Criteria:

* Diagnosis of poor prognosis advanced cancer defined as locally advanced or metastatic cancer (e.g., pancreaticobiliary, esophagogastric, hepatocellular carcinoma, lung, or gynecological cancer) and/or disease progression following at least first line chemotherapy.
* Ability to provide informed consent
* Identification of an informal caregiver
* Oncologist reported discussion of prognosis with the patient and/or caregiver.

Patient Exclusion Criteria:

* Not fluent in English
* Severely cognitively impaired (as measured by Short Portable Mental Status Questionnaire scores of < 6)
* Too ill or weak to complete the interviews (as judged by the interviewer)
* Currently receiving palliative care/hospice at the time of enrollment
* Children and young adults under age 18
* Deemed inappropriate for the study by their treating oncologist.
* In addition, patient-caregiver dyads in which both members have an accurate understanding of prognosis (terminal status and life-expectancy) will be excluded due to the lack of need for an intervention.

Caregiver inclusion criteria:

* The person (family member or friend) whom the patient indicates provides their informal (unpaid) care
* English speaking
* Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan J Shen, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Started | 14 | 14
Completed | 8 (*Note: Whereas 8 patients completed the study, 1 additional patient was able to be included in the analysis of most patient outcome measures as they completed the applicable assessments for those measures prior to being lost to follow-up.) | 8
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.36 (9.27) | 57.07 (13.38) | 58.21 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed for caregivers' sex (n=13) differs from total sample (n=14) because one caregiver refused to designate sex/gender.
  Participants
    number analyzed (Participants) | 14 | 13 | 27
    Female | 8 | 7 | 15
    Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Prognostic Understanding
Description: Change in prognostic understanding is assessed at baseline and post-intervention with two items on prognostic understanding: (1) Terminal illness acknowledgement with the item "How would you describe your current health status?" Answer choices include: 1) Relatively healthy, 2) relatively healthy but terminally ill, 3) seriously ill but not terminally ill, and 4) seriously ill and terminally ill, and (5) I don't know]. Responses 2 and 4 are coded as accurate and responses 1, 3, and 5 are coded as inaccurate. (2) Life-expectancy [Months, Years, and "I don't know"]. Months are coded as accurate and years and I don't know are coded as inaccurate. Each variable is coded as 0=inaccurate or 1=accurate, for a total summary score range of 0 to 2. Differences between baseline and post-intervention assessments are calculated (possible range, -2 to +2) to determine changes in prognostic understanding.
Time Frame: Baseline, post-intervention (within 30 days)
Population: The number of patients analyzed (n=9) was less than the total patients enrolled (n=14) because n=3 patients withdrew from the study and n=2 patients were lost to follow up and did not have post-intervention data. The number of caregivers analyzed (n=8) was less than the total caregivers enrolled (n=14) because n=3 caregivers withdrew from the study and n=3 were lost to follow up and did not have post-intervention data.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 9 | 8
Change in scores on a scale | 0.00 (0.50) | 0.25 (0.46)

2. Secondary Outcome: Change in Patients' Engagement in Advance Care Planning, as Measured by the Decision Maker Subscale of the Advance Care Planning Engagement Survey: Action Measures, From Baseline to Post-intervention
Description: Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Decision Maker (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options include: yes=1, no=0. Questions include those asking about whether patients have engaged in a decision around advance care planning (e.g., "Have you already decided who you want your medical decision maker to be?" Individual scores can range from 0 to 4, with higher scores indicating that more decisions have been made around advance care planning. Change scores can range from -4 to +4.
Time Frame: Baseline, post-intervention (within 30 days)
Population: There are n=0 caregivers for this measure because this outcome variable was only assessed among patients. The number of patients analyzed (n=9) was less than the total patients enrolled (n=14) because n=3 patients withdrew from the study and n=2 patients were lost to follow up and did not have post-intervention data.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 9 | 0
Change in scores on a scale | 0.44 (1.24) |

3. Secondary Outcome: Change in Patients' Engagement in Advance Care Planning, as Measured by the Decision Maker Subscale of the Advance Care Planning Engagement Survey: Action Measures, From Baseline to 3-month Follow-up
Description: as for outcome 2
Time Frame: Baseline, follow-up (3 months)
Population: There are n=0 caregivers for this measure because this outcome variable was only assessed among patients. The number of patients analyzed (n=7) was less than the total patients enrolled (n=14) because n=3 patients withdrew from the study, n=3 patients were lost to follow up and did not have post-intervention data, and n=1 patient did not provide data for this measure.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 7 | 0
Change in scores on a scale | 1.14 (1.21) |

4. Secondary Outcome: Change in Patients' Engagement in Advance Care Planning, as Measured by the Quality of Life Subscale of the Advance Care Planning Engagement Survey: Action Measures, From Baseline to Post-intervention
Description: Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Quality of Life (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options include: yes=1, no=0. Questions include those asking about whether patients have engaged in a decision around quality of life in advance care planning (e.g., "Have you already decided whether or not certain health situations would make your life not worth living?" Individual scores can range from 0 to 4, with higher scores indicating that more decisions have been made around advance care planning as it pertains to quality of life. Change scores can range from -4 to +4.
Time Frame: Baseline, post-intervention (within 30 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 9 | 0
Change in scores on a scale | 0.78 (1.09) |

5. Secondary Outcome: Change in Patients' Engagement in Advance Care Planning, as Measured by the Quality of Life Subscale of the Advance Care Planning Engagement Survey: Action Measures, From Baseline to 3-month Follow-up
Description: as for outcome 4
Time Frame: Baseline, follow-up (3 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 7 | 0
Change in scores on a scale | 0.57 (0.96) |

6. Secondary Outcome: Change in Caregivers' Engagement in Advance Care Planning, as Measured by the Van Scoy and Sudore Measure Which Adapts the Decision Maker Subscale of the Advance Care Planning Engagement Survey, From Baseline to Post-Intervention
Description: Change in caregiver engagement in advance care planning will be assessed with a companion measure in the final phases of validation by Van Scoy and Sudore. This measure adapts the Advance Care Planning Engagement Survey to apply to caregivers. Response options include: yes=1, no=0. Individual scores can range from 0 to 4, with higher scores indicating more decisions have been made. Change scores can range from -4 to +4.
Time Frame: Baseline, post-intervention (within 30 days)
Population: There are n=0 patients for this measure because this outcome variable was only assessed among caregivers. The number of caregivers analyzed (n=8) was less than the total caregivers enrolled (n=14) because n=3 caregivers withdrew from the study and n=3 were lost to follow up and did not have post-intervention data.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 0 | 8
Change in scores on a scale |  | -0.50 (0.93)

7. Secondary Outcome: Change in Caregivers' Engagement in Advance Care Planning, as Measured by the Van Scoy and Sudore Measure Which Adapts the Decision Maker Subscale of the Advance Care Planning Engagement Survey, From Baseline to 3-month Follow-up
Description: as for outcome 6
Time Frame: Baseline, follow-up (3 months)
Population: There are n=0 patients for this measure because this outcome variable was only assessed among caregivers. The number of caregivers analyzed (n=7) was less than the total caregivers enrolled (n=14) because n=3 caregivers withdrew from the study, n=3 were lost to follow up and did not have post-intervention data, and n=1 did not provide data for this outcome.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 0 | 7
Change in scores on a scale |  | .14 (1.57)

8. Secondary Outcome: Change in the Number of Advance Directives Completed
Description: Completion of advance directives will be assessed by asking patients whether they completed a do-not-resuscitate order, a living will, and/or identified a health care proxy; data will be verified through the patient's electronic health record. Change in these numbers will be assessed at baseline and post-intervention. Scores are computed by summing together the total number of advance directives completed. Scores can range from 0 to 3, with higher scores indicating increases in completion of advance directives. Change scores can range from -3 to +3.
Time Frame: Baseline, post-intervention (within 30 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in completed advance directives
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 9 | 0
Change in completed advance directives | 0.56 (1.01) |

9. Secondary Outcome: Change in Psychological Distress, as Measured by the Hospital Anxiety and Depression Scale (HADS)
Description: Psychological distress will be measured using the Hospital Anxiety and Depression Scale (HADS), a valid and reliable 14-item, Likert-type self-report measure of mood disturbance commonly used with cancer patients. The HADS contains two seven-item subscales: 1) anxiety and 2) depressive symptoms. Each item on this scale is rated on a 4-point scale (0 to 3), and all items are summed to create a HADS total score. Total scores can range from 0 to 42, with higher numbers indicating higher levels of distress. Change in psychological distress will be assessed at baseline and post-intervention.
Time Frame: Baseline, post-intervention (within 30 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 9 | 8
Change in scores on a scale | 0.33 (6.54) | -2.12 (5.79)

10. Secondary Outcome: Change in Communication Quality, as Measured by the Family Communication Subscale of the Cancer Communication Assessment Tool for Patients and Families (CCAT-PF)
Description: Communication quality will be assessed with the 5-item Family Communication subscale of the Cancer Communication Assessment Tool for Patients and Families, a valid measure in cancer patients and caregivers. Response options are on a 5-point Likert-type scale (1 = strongly disagree to 5= strongly agree). Scores can range from 5 to 25, with higher scores indicating worse communication quality. Change in communication quality will be assessed at baseline and post-intervention.
Time Frame: Baseline, post-intervention (within 30 days)
Population: The original CCAT scale is scored on a scale from 1 to 6, but this data had a 1 to 5 response scale. The number of patients analyzed (n=9) was less than the total patients enrolled (n=14) because n=3 patients withdrew from the study and n=2 patients were lost to follow up. The number of caregivers analyzed (n=8) was less than the total caregivers enrolled (n=14) because n=3 caregivers withdrew from the study and n=3 were lost to follow up.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 9 | 8
Change in scores on a scale | -1.33 (6.63) | 0.50 (2.00)

11. Secondary Outcome: Change in Caregiver Burden (Caregivers Only), as Measured by the Zarit Burden Interview
Description: Caregiver burden will be assessed with the Zarit Burden Interview (ZBI), a reliable and valid 22-item measure of caregiver burden used in intervention studies of cancer caregivers. Response options are on a 5-point Likert-type scale (0 = never to 4=nearly always). Scores can range from 0 to 88, with higher scores indicating higher levels of burden. Change in caregiver burden will be assessed at baseline and post-intervention.
Time Frame: Baseline, post-intervention (within 30 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
Number analyzed (Participants) | 0 | 8
Change in scores on a scale |  | -4.13 (9.00)

ADVERSE EVENTS:
Time Frame: 3 months (during study period)
Arm/Group | Patient Intervention Arm | Caregiver (of Patient) Intervention Arm
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
The statistical analysis plan (and associated statistical power) was based on an expected sample size of 30 evaluable dyads. Due to COVID-19 and restrictions around data collection, only 14 dyads were consented and 8 dyads were evaluable (with n=9 patients, n=8 caregivers). This reduced sample size was not sufficient for the statistical analysis plan as written, and, therefore, only descriptive statistics for the response proportions can be presented for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT03833817/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03833817/ICF_001.pdf